CLINICAL TRIAL: NCT07009314
Title: Scaling Out S.A.F.E. Firearm Across Two Health Systems as a Universal Suicide Prevention Strategy (SCALE ASPIRE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Henry Ford Health System (Other); Kaiser Permanente (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AWD00002547; R01MH138333 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Suicide
Keywords: implementation science; firearms; suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized controlled trial
Masking Description: Data analyst and biostatistician will be blinded to randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Implementation phase (training, EHR nudge, and facilitation received; S.A.F.E. Firearm delivered) (Experimental): Each group of clinics will cross over from the baseline phase to the implementation phase, one at a time. In the implementation phase, the implementation approaches (training, EHR nudge, facilitation) and the S.A.F.E. Firearm program will be implemented. S.A.F.E. Firearm consists of health care staff having a secure firearm storage discussion with a patient during their visit and offering them a free cable firearm lock. The implementation phase will last for 6 months for each group of clinics.
  Interventions: Behavioral: Implementation package (training, facilitation, electronic health record nudge)
- Baseline data collection phase (usual care) (No Intervention): The study will begin with a baseline data collection phase. During the baseline data collection phase, no clinics will be exposed to S.A.F.E. Firearm nor the implementation approaches (training, EHR nudge, facilitation). The length of the baseline data collection phase will differ between each "wedge" (i.e., group of clinics) depending on when the group is randomly assigned to cross over into the implementation phase. All clinics will be in the baseline data collection phase for at least six months before the interventions are activated.
- Maintenance phase (training and facilitation removed) (No Intervention): After the six-month period during which the implementation strategies (training, EHR nudge, facilitation) are enacted at a clinic, the research team will assess outcomes during the remainder of the study period in a "maintenance" phase.
  No additional training or facilitation will be received during this maintenance period following the implementation period. Clinics will still receive ongoing data reports, the the EHR nudge will remain turned on, and clinics will continue to deliver the S.A.F.E. Firearm program.

INTERVENTIONS:
Behavioral: Implementation package (training, facilitation, electronic health record nudge) — Training will consist of an initial presentation on S.A.F.E. Firearm by the study team, informational resources to support program delivery, and recommendations for self-guided continuing medical education programs.
  Facilitation will last 6 months at each site. It may involve 1) a readiness assessment for each clinic to identify implementation barriers and develop relationships with constituents; 2) kick-off meetings at trial launch, at which staff will identify how to implement S.A.F.E. Firearm in the clinic; 3) goal-setting within the first few months of the program; 4) trouble-shooting to address barriers identified during the pre-implementation readiness assessment and emergent challenges; and 5) designing a sustainment plan to maintain the program for future years.
  A clinician decision support ("nudge"), designed to align with best practices within each health system, will be deployed in the EHR workflow to remind clinicians to deliver S.A.F.E. Firearm and offer a cable lock.
  Arms: Implementation phase (training, EHR nudge, and facilitation received; S.A.F.E. Firearm delivered)

SUMMARY:
In this randomized controlled trial, researchers will assess the expansion of the S.A.F.E. Firearm program into adult primary care and women's health at two health systems in Michigan and Colorado that have previously implemented S.A.F.E. Firearm in pediatrics. S.A.F.E. Firearm involves a brief conversation between health care staff and patients about secure firearm storage and an offer of a free firearm cable lock. Researchers will test S.A.F.E. Firearm and a package of strategies intended to help health care staff incorporate the program into their practice. The strategies include: training, a prompt in the electronic health record, and facilitation, or tailored problem-solving support.

The study seeks to answer the following questions:

* How effective is S.A.F.E. Firearm at changing patients' firearm storage behavior?
* How effective is the implementation strategy package at increasing delivery of the S.A.F.E. Firearm program?

Some patients and health care staff will be invited to participate in surveys and/or interviews about their experiences with S.A.F.E. Firearm and the implementation strategy package.

DETAILED DESCRIPTION:
Reducing unauthorized access to firearms is a population-level suicide prevention strategy. S.A.F.E. Firearm is a universal evidence-based suicide prevention intervention primed for implementation nationally. In the largest hybrid type III effectiveness-implementation trial of its kind, funded by the National Institute of Mental Health (NIMH; "ASPIRE" trial), we tested how to implement S.A.F.E. Firearm across approximately 45,000 well-child visits in 30 pediatric primary care clinics at Henry Ford Health (HFH) in Michigan and Kaiser Permanente Colorado (KPCO). We found that training, an electronic health record (EHR)-based clinician decision support ("nudge"), and facilitation (i.e., implementation support to clinics) resulted in robust practice change from approximately 2% reach (baseline) to 49% reach (active implementation). While the ASPIRE trial focused on delivery of the intervention to parents of young people, we have the rare opportunity to expand S.A.F.E. Firearm delivery for all adults via adult primary care and women's health clinics, offering a new context and broadened population. This holds promise given that (a) many of these patients will have children in their homes (e.g., parents, grandparents) and (b) adults may benefit from S.A.F.E. Firearm themselves because putting time and space between adults and loaded firearms can reduce firearm suicide.

The proposed study ("SCALE-ASPIRE") is motivated by HFH and KPCO constituents' eagerness to implement this intervention beyond pediatric primary care and will advance the science of implementation by understanding how to "scale-out" successful intervention and implementation efforts. In SCALE-ASPIRE, we will conduct a stepped wedge cluster randomized hybrid type II effectiveness-implementation trial in approximately 48 clinics in adult primary care and women's health at HFH and KPCO. In Aim 1, in collaboration with key partners including clinicians, leaders, and patients, we will use the ADAPT-ITT approach to adapt S.A.F.E. Firearm for the new clinic context and broadened population. In Aim 2, we will test the effectiveness of S.A.F.E. Firearm and our implementation approach (training, EHR nudge, facilitation) on effectiveness (firearm storage behavior, co-primary; suicide attempts, suicide deaths, and all-cause firearm injury and mortality in adults and young people, secondary) and implementation (reach, or patient-reported receipt of S.A.F.E. Firearm, co-primary; implementation fidelity and cost, secondary) outcomes. In Aim 3, we will use mixed methods to elucidate intervention and implementation mechanisms and to better understand heterogeneity across levels. Specifically, we will conduct interviews to understand constituent perspectives, and explore how patient, clinician, and clinic factors relate to heterogeneity in our co-primary outcomes. Study results will guide the identification of effective secure firearm storage interventions, increase knowledge of effective implementation strategies in large health systems, and advance the literature on scaling out successful intervention and implementation efforts to new populations and settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18+ years of age and attend an eligible visit within a participating specialty (adult primary care, women's health) at a participating clinic within the Henry Ford Health or Kaiser Permanente Colorado health systems
* Health care personnel must be 18+ years of age and employed by a participating health care clinic within the Henry Ford Health or Kaiser Permanente Colorado health systems

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5442 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Firearm storage behavior | Firearm storage behavior will be collected via survey sent to patients after visits for the 3-year study period (baseline through maintenance phases)
  Patients who indicate that there are firearms in or around their homes will be asked to report their firearm storage practices in (a) the 2 weeks prior to the visit; and (b) the 2 weeks after the visit. Respondents will indicate whether none, some, or all firearms were stored locked at each time point. Locked storage refers to storage in a container that limits access to the firearm (e.g., safe, cabinet, case) and/or storage with a cable or trigger lock.
Patient-reported reach of the S.A.F.E. Firearm program | Reach will be collected via survey sent to patients after visits for the 3-year study period (baseline through maintenance phases)
  The proportion of eligible visits for which patients report receiving the two components of S.A.F.E. Firearm (discussion of secure firearm storage, offer of a free cable firearm lock)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kaiser Permanente Colorado, Aurora, Colorado
  - Henry Ford Health, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Undecided